## Prueba T

| | Notas | |
|---|---|---|
| Results | | 6/15/2017 18:51 |
| Comments | | |
| Intput | Data | C:\Users\carlo\Desktop\Ca |
| | Active data set<br>Filter<br>Weight | Conjunto_de_datos1 <none></none> |
| | Row | <none></none> |
| | No. Rows file | <none></none> |
| | No. Rows file | 100 |
| Treatment of lost values | Definition of lost values | The lost values defined by the user will be treated as lost |
| | Cases used | The statistics of each analysis are based on cases that do not have lost data or are out of range in any of the variables of the analysis. |
| Sintax | | T-TEST GROUPS=CasosvsContro les(1 2) /MISSING=ANALYSIS /VARIABLES=P01 P02 P03 P04 P05 P06 P07 P08 P09 P10 P11 P12 P13 P14 P15 P16 P17 P18 P19 P20 /CRITERIA=CI(.95). |
| Resources | Processor time | 00:00:00,00 |
| | Time elapsed | 00:00:00,01 |

[Data\_set1] C:\Users\carlo\Desktop\Casos y Controles.sav

## Group statistics

| | 0.0up 0.u | | | | |
|---|---|---|---|---|---|
| | | | | Typical | Typical |
| Cases Vs Controls | | N | Mean | deviation | error |
| Age in years | Cases | 50 | 44.60 | 13.368 | 1.890 |
| | Controls | 50 | 65.22 | 11.915 | 1.685 |
| Edad | Cases | 50 | 3.50 | 1.329 | 0.188 |
| 1 | Controls | 50 | 5.56 | 1.248 | 0.176 |
| Age of UI symptom | Cases | 50 | 1.76 | 0.431 | 0.061 |
| | Controls | 50 | 1.88 | 0.328 | 0.046 |
| Urinary incontinence | Cases | 28 | 3.21 | 0.876 | 0.166 |
| | Controls | 50 | 3.44 | 0.884 | 0.125 |
| Urgency | Cases | 50 | 1.30 | 0.463 | 0.065 |
| | Controls | 50 | 1.04 | 0.198 | 0.028 |
| Increased Daytime frequency | Cases | 50 | 1.40 | 0.495 | 0.070 |
| | Controls | 50 | 1.16 | 0.370 | 0.052 |
| Nocturia | Cases | 50 | 1.40 | 0.495 | 0.070 |
| | Controls | 50 | 1.36 | 0.485 | 0.069 |
| Nocturnal enuresis | Cases | 50 | 1.96 | 0.198 | 0.028 |
| | Controls | 50 | 1.84 | 0.370 | 0.052 |
| Pelvic pain | Cases | 50 | 1.48 | 0.505 | 0.071 |
| | Controls | 50 | 2.00 | 0.000 | 0.000 |
| Feeling of POP | Cases | 50 | 1.50 | 0.735 | 0.104 |
| | Controls | 50 | 1.70 | 0.463 | 0.065 |
| UTIs | Cases | 50 | 1.78 | 0.418 | 0.059 |
| | Controls | 50 | 1.96 | 0.198 | 0.028 |
| Constipation | Cases | 50 | 1.90 | 0.303 | 0.043 |
| | Controls | 50 | 1.46 | 0.503 | 0.071 |
| Feeling of incomplete emtiying | Cases | 50 | 1.24 | 0.431 | 0.061 |
| | Controls | 50 | 1.62 | 0.490 | 0.069 |
| Disuria | Cases | 50 | 1.48 | 0.505 | 0.071 |
| | Controls | 50 | 1.62 | 0.490 | 0.069 |
| LUTs | Cases | 50 | 1.48 | 0.735 | 0.104 |
| | Controls | 50 | 0.46 | 0.646 | 0.091 |
| Overactive bladder | Cases | 50 | 1.76 | 0.431 | 0.061 |
| | Controls | 50 | 1.48 | 0.505 | 0.071 |
| Stress UI | Cases | 50 | 1.90 | 0.303 | 0.043 |
| ** | Controls | 50 | 1.58 | 0.499 | 0.071 |
| Increased bladder sensation | Cases | 50 | 1.86 | 0.351 | 0.050 |
| | Controls | 50 | 1.80 | 0.404 | 0.057 |
| | | - 00 | 00 | 504 | 0.001 |

| Obstruction | Cases | 50 | 1.98 | 0.141 | 0.020 |
|-------------|----------|----|------|-------|-------|
| | Controls | 50 | 1.78 | 0.418 | 0.059 |
| Flowmetry | Cases | 50 | 0.16 | 0.468 | 0.066 |
| | Controls | 50 | 0.94 | 1.077 | 0.152 |

## Independent samples test

| Independent samples test | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| 1 | | Levene's test for equality of | f variances | | | Test T for equality of means | | | ı | |
| | | | | | | | | inte | | 95% Confidence<br>interval for the<br>difference |
| | | F | Sig. | t | gl | Sig.<br>(bilateral) | Difference of means | error of the<br>difference | lower | higher |
| Age in years | Equal variances have been | 1.190 | 0.278 | -8.142 | 98 | 0.000 | -20.620 | 2.532 | -25.646 | -15.594 |
| | No equal variances have been assumed | | | -8.142 | 96.731 | 0.000 | -20.620 | 2.532 | -25.646 | -15.594 |
| Edad | Equal variances have been | 0.418 | 0.519 | -7.991 | 98 | 0.000 | -2.060 | 0.258 | -2.572 | -1.548 |
| | No equal variances have been assumed | | | -7.991 | 97.618 | 0.000 | -2.060 | 0.258 | -2.572 | -1.548 |
| Age of UI symptom | Equal variances have been | 10.480 | 0.002 | -1.565 | 98 | 0.121 | -0.120 | 0.077 | -0.272 | 0.032 |
| | No equal variances have been assumed | | | -1.565 | 91.494 | 0.121 | -0.120 | 0.077 | -0.272 | 0.032 |
| Urinary incontinence | Equal variances have been | 0.000 | 0.985 | -1.085 | 76 | 0.281 | -0.226 | 0.208 | -0.640 | 0.189 |
| | No equal variances have been assumed | | | -1.088 | 56.482 | 0.281 | -0.226 | 0.207 | -0.641 | 0.190 |
| Urgency | Equal variances have been | 87.313 | 0.000 | 3.652 | 98 | 0.000 | 0.260 | 0.071 | 0.119 | 0.401 |
| | No equal variances have been assumed | | | 3.652 | 66.340 | 0.001 | 0.260 | 0.071 | 0.118 | 0.402 |
| Increased Daytime frequency | Equal variances have been | 30.464 | 0.000 | 2.746 | 98 | 0.007 | 0.240 | 0.087 | 0.067 | 0.413 |
| | No equal variances have been assumed | | | 2.746 | 90.778 | 0.007 | 0.240 | 0.087 | 0.066 | 0.414 |
| Nocturia | Equal variances have been | 0.653 | 0.421 | 0.408 | 98 | 0.684 | 0.040 | 0.098 | -0.154 | 0.234 |
| | No equal variances have been assumed | | | 0.408 | 97.959 | 0.684 | 0.040 | 0.098 | -0.154 | 0.234 |
| Nocturnal enuresis | Equal variances have been | 19.085 | 0.000 | 2.021 | 98 | 0.046 | 0.120 | 0.059 | 0.002 | 0.238 |
| | No equal variances have been assumed | | | 2.021 | 74.887 | 0.047 | 0.120 | 0.059 | 0.002 | 0.238 |
| Pelvic pain | Equal variances have been | 30576.000 | 0.000 | -7.286 | 98 | 0.000 | -0.520 | 0.071 | -0.662 | -0.378 |
| | No equal variances have been assumed | | | -7.286 | 49.000 | 0.000 | -0.520 | 0.071 | -0.663 | -0.377 |
| Feeling of POP | Equal variances have been | 15.400 | 0.000 | -1.627 | 98 | 0.107 | -0.200 | 0.123 | -0.444 | 0.044 |
| | No equal variances have been assumed | | | -1.627 | 82.561 | 0.107 | -0.200 | 0.123 | -0.444 | 0.044 |
| UTIs | Equal variances have been | 40.288 | 0.000 | -2.750 | 98 | 0.007 | -0.180 | 0.065 | -0.310 | -0.050 |
| | No equal variances have been assumed | | | -2.750 | 69.884 | 0.008 | -0.180 | 0.065 | -0.311 | -0.049 |
| Constipation | Equal variances have been | 83.084 | 0.000 | 5.295 | 98 | 0.000 | 0.440 | 0.083 | 0.275 | 0.605 |
| | No equal variances have been assumed | | | 5.295 | 80.387 | 0.000 | 0.440 | 0.083 | 0.275 | 0.605 |
| Feeling of incomplete emtiying | Equal variances have been | 8.820 | 0.004 | -4.114 | 98 | 0.000 | -0.380 | 0.092 | -0.563 | -0.197 |
| | No equal variances have been assumed | | | -4.114 | 96.438 | 0.000 | -0.380 | 0.092 | -0.563 | -0.197 |
| Disuria | Equal variances have been | 2.750 | 0.100 | -1.407 | 98 | 0.163 | -0.140 | 0.100 | -0.337 | 0.057 |
| | No equal variances have been assumed | | | -1.407 | 97.918 | 0.163 | -0.140 | 0.100 | -0.337 | 0.057 |
| LUTs | Equal variances have been | 1.378 | 0.243 | 7.372 | 98 | 0.000 | 1.020 | 0.138 | 0.745 | 1.295 |
| | No equal variances have been assumed | | | 7.372 | 96.391 | 0.000 | 1.020 | 0.138 | 0.745 | 1.295 |
| Overactive bladder | Equal variances have been | 17.802 | 0.000 | 2.982 | 98 | 0.004 | 0.280 | 0.094 | 0.094 | 0.466 |
| | No equal variances have been assumed | | | 2.982 | 95.685 | 0.004 | 0.280 | 0.094 | 0.094 | 0.466 |
| Stress UI | Equal variances have been | 72.439 | 0.000 | 3.878 | 98 | 0.000 | 0.320 | 0.083 | 0.156 | 0.484 |
| | No equal variances have been assumed | | | 3.878 | 80.858 | 0.000 | 0.320 | 0.083 | 0.156 | 0.484 |
| Increased bladder sensation | Equal variances have been | 2.561 | 0.113 | 0.793 | 98 | 0.430 | 0.060 | 0.076 | -0.090 | 0.210 |
| | No equal variances have been assumed | | | 0.793 | 96.084 | 0.430 | | | | |
| Obstruction | Equal variances have been | 63.002 | 0.000 | 3.202 | 98 | 0.002 | 0.200 | 0.062 | 0.076 | 0.324 |
| | No equal variances have been assumed | | | 3.202 | 60.049 | 0.002 | | | 0.075 | |
| Flowmetry | Equal variances have been | 24.839 | 0.000 | -4.698 | 98 | 0.000 | -0.780 | 0.166 | -1.109 | -0.451 |
| | No equal variances have been assumed | | | -4.698 | 66.854 | 0.000 | | | | -0.449 |
| | | | | | | | l . | | l | |